CLINICAL TRIAL: NCT02054741
Title: A Geriatric Assessment Intervention for Patients Aged 70 and Over Receiving Chemotherapy or Similar Agents for Advanced Cancer: Reducing Toxicity in Older Adults
Brief Title: Geriatric Assessment Intervention for Reducing Toxicity in Older Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supriya Mohile (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Chicago (Other); City of Hope National Medical Center (Other)
Responsible Party: Sponsor-Investigator, Supriya Mohile, Professor, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: URCC13059; NCI-2013-01904 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC13059 (Other: University of Rochester); URCC-13059 (Other: DCP); URCC-13059 (Other: CTEP); UG1CA189961 (NIH); U10CA037420 (NIH); R01CA177592 (NIH); NCT02066168 (obsolete NCT alias)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Adult Solid Neoplasm; Toxicity; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (GA intervention) (Experimental): Patients complete a geriatric assessment. Patients and physicians are provided with the geriatric assessment information and recommendations.
  Interventions: Other: Comprehensive Geriatric Assessment; Other: Quality-of-Life Assessment; Other: Survey Administration
- Arm II (usual care) (No Intervention): Patients complete a geriatric assessment, but information other than clinically significant cognitive impairment and depression is not provided to the oncology teams.

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Complete geriatric assessment
  Other Names: geriatric assessment
  Arms: Arm I (GA intervention)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm I (GA intervention)
Other: Survey Administration — Ancillary studies
  Arms: Arm I (GA intervention)

SUMMARY:
This cluster randomized clinical trial compares a geriatric assessment intervention with usual care for reducing cancer treatment toxicity in older patients with cancer that has spread to other places in the body. A geriatric assessment may identify risk factors for cancer treatment toxicity and may improve outcomes for older patients with advanced cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if providing information regarding geriatric assessment (GA) and GA-driven recommendations to oncology physicians reduces clinician-rated grade 3-5 toxicity in patients aged 70 and over with advanced cancer starting a new treatment regimen.

SECONDARY OBJECTIVES:

I. Proportion of patients who are alive at 6 months after study entry. II. Evaluate whether providing oncology physicians with information regarding GA summary and GA-driven recommendations influences clinical care of older patients receiving treatment for advanced cancer.

IIA. Compare treatment decisions (as measured by relative dose intensity of the agents administered in the first cycle).

IIB. Describe the number and type of GA-driven recommendations implemented for older patients starting a new treatment regimen for advanced cancer.

OUTLINE: Treatment sites are randomized to 1 of 2 arms.

ARM I (GA intervention): Patients complete a geriatric assessment. Patients and physicians are provided with the geriatric assessment information and recommendations.

ARM II (usual care): Patients complete a geriatric assessment, but information other than clinically significant cognitive impairment and depression is not provided to the oncology teams.

After completion of study, patients are followed up at 4-6 weeks, at 3 and 6 months, and at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR PHYSICIANS
* Oncology physicians must work at a National Cancer Institute (NCI) Community Oncology Research Program (NCORP) practice site with no plans to leave that NCORP practice site or retire at the time of enrollment into the study
* INCLUSION CRITERIA FOR PATIENTS
* Diagnosis of an advanced solid tumor malignancy (advanced cancer) or lymphoma; in most situations, this would be a stage IV cancer; patients with a diagnosis of stage III cancer or lymphoma are eligible if cure is not possible or anticipated; clinical staging without pathological confirmation of advanced disease is allowed
* Plan to start a new cancer treatment regimen within 4 weeks from time of baseline registration; the treatment regimen is up to the discretion of the treating oncology physician; the regimen must include a chemotherapy drug or other agents that have similar prevalence of toxicity; patients who will receive monoclonal antibody therapy or other cancer therapies (e.g., tyrosine kinase inhibitors) are eligible if other agents present a prevalence of toxicity similar to chemotherapy; patients who are receiving approved cancer treatment in combination with radiation are eligible; a patient may also be enrolled on a treatment trial and participate in this study, if all other inclusion and exclusion criteria are met. *Chemotherapy is defined as cytotoxic drugs; in addition, agents (e.g., monoclonal antibodies and targeted agents) that have a prevalence of grade 3-5 toxicity in older patients similar to chemotherapy (>50%) will be allowed.
* Plan to be on chemotherapy or other allowable treatment for at least 3 months (minimum 70 days) and be willing to come in for study visits
* Have at least one geriatric assessment domain meet the cut-off score for impairment other than polypharmacy
* Able to provide informed consent, or if the oncology physician determines the patient to not have decision-making capacity, a patient-designated health care proxy (or authorized representative per institutional policies) must sign consent by the baseline visit. If the participant is found to be impaired on the Blessed-Orientation Memory Concentration Test (BOMC) during screening; they must have a health care proxy or authorized representative to be eligible to enroll.
* Participant has adequate understanding of the English language

Exclusion Criteria:

* EXCLUSION CRITERIA FOR PATIENTS
* Have surgery planned within 3 months of consent; patients who have previously received surgery are eligible
* Presence of symptomatic brain metastases at time of study consent process. Patients with a history of treated brain metastases are eligible if they are not symptomatic at the time of study enrollment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 733 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Mohile, Principal Investigator — University of Rochester NCORP Research Base
Locations (23):
- United States (23):
  - City of Hope, Duarte, California
  - Delaware/Christiana Care NCORP, Newark, Delaware
  - Hawaii MU-NCORP, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Heartland NCORP, Decatur, Illinois
  - Kansas City NCORP, Prairie Village, Kansas
  - Wichita NCORP, Wichita, Kansas
  - Gulf South MU-NCORP, New Orleans, Louisiana
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Metro Minnesota NCORP, Minneapolis, Minnesota
  - Kansas City NCORP, Kansas City, Missouri
  - Nevada NCORP, Las Vegas, Nevada
  - North Shore LIJ Health System NCORP, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Southeast Clinical Oncology Research Program, Winston-Salem, North Carolina
  - Columbus NCORP, Columbus, Ohio
  - Dayton NCORP, Dayton, Ohio
  - Pacific Cancer Research Consortium Ncorp, Portland, Oregon
  - Geisinger Cancer Institute NCORP, Danville, Pennsylvania
  - NCORP of the Carolinas, Greenville, South Carolina
  - Northwest NCORP, Tacoma, Washington
  - Wisconsin NCORP, Marshfield, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Flannery MA, Zhang Z, Culakova E, Loh KP, Canin B, Tylock RG, Stauffer FA, Mohamed M, Sun H, Mohile S. Decision regret in older adults with advanced cancer receiving systemic therapy: Associations with patient-reported and clinician-rated tolerability metrics. Cancer. 2025 Oct 15;131 Suppl 2(Suppl 2):e70023. doi: 10.1002/cncr.70023. PMID 41123568
- [Derived] Mohamed MR, Juba K, Awad H, Flannery M, Culakova E, Wells M, Cacciatore J, Jensen-Battaglia M, Mohile S, Ramsdale E. Effect of polypharmacy and potentially inappropriate medications on physical functional decline among older adults with advanced cancer receiving systemic treatment. Support Care Cancer. 2024 Sep 19;32(10):674. doi: 10.1007/s00520-024-08877-6. PMID 39294452
- [Derived] Lund JL, Cacciatore J, Tylock R, Su IH, Sharma S, Hinton SP, Smith S, Nowels MA, Chen X, Duberstein PR, Hanson LC, Mohile SG. Development and Evaluation of a Multisource Approach to Extend Mortality Follow-Up for Older Adults With Advanced Cancer Enrolled in Randomized Trials. JCO Clin Cancer Inform. 2024 Apr;8:e2300183. doi: 10.1200/CCI.23.00183. PMID 38564692
- [Derived] Ramsdale E, Kunduru M, Smith L, Culakova E, Shen J, Meng S, Zand M, Anand A. Supervised learning applied to classifying fallers versus non-fallers among older adults with cancer. J Geriatr Oncol. 2023 May;14(4):101498. doi: 10.1016/j.jgo.2023.101498. Epub 2023 Apr 19. PMID 37084629
- [Derived] Xu H, Mohamed M, Flannery M, Peppone L, Ramsdale E, Loh KP, Wells M, Jamieson L, Vogel VG, Hall BA, Mustian K, Mohile S, Culakova E. An Unsupervised Machine Learning Approach to Evaluating the Association of Symptom Clusters With Adverse Outcomes Among Older Adults With Advanced Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e234198. doi: 10.1001/jamanetworkopen.2023.4198. PMID 36947036
- [Derived] Mohamed MR, Loh KP, Mohile SG, Sohn M, Webb T, Wells M, Yilmaz S, Tylock R, Culakova E, Magnuson A, Sun CL, Bearden J, Hopkins JO, Faller BA, Klepin HD. External Validation of Risk Factors for Unplanned Hospitalization in Older Adults With Advanced Cancer Receiving Chemotherapy. J Natl Compr Canc Netw. 2023 Mar;21(3):273-280.e3. doi: 10.6004/jnccn.2022.7094. PMID 36898361
- [Derived] Mohamed MR, Mohile SG, Juba KM, Awad H, Wells M, Loh KP, Flannery M, Culakova E, Tylock RG, Ramsdale EE. Association of polypharmacy and potential drug-drug interactions with adverse treatment outcomes in older adults with advanced cancer. Cancer. 2023 Apr 1;129(7):1096-1104. doi: 10.1002/cncr.34642. Epub 2023 Jan 24. PMID 36692475
- [Derived] Culakova E, Mohile SG, Peppone L, Ramsdale E, Mohamed M, Xu H, Wells M, Tylock R, Java J, Loh KP, Magnuson A, Jamieson L, Vogel V, Duberstein PR, Chapman BP, Dale W, Flannery MA. Effects of a Geriatric Assessment Intervention on Patient-Reported Symptomatic Toxicity in Older Adults With Advanced Cancer. J Clin Oncol. 2023 Feb 1;41(4):835-846. doi: 10.1200/JCO.22.00738. Epub 2022 Nov 10. PMID 36356279
- [Derived] Presley CJ, Mohamed MR, Culakova E, Flannery M, Vibhakar PH, Hoyd R, Amini A, VanderWalde N, Wong ML, Tsubata Y, Spakowicz DJ, Mohile SG. A Geriatric Assessment Intervention to Reduce Treatment Toxicity Among Older Adults With Advanced Lung Cancer: A Subgroup Analysis From a Cluster Randomized Controlled Trial. Front Oncol. 2022 Mar 31;12:835582. doi: 10.3389/fonc.2022.835582. eCollection 2022. PMID 35433441
- [Derived] Mohile SG, Mohamed MR, Xu H, Culakova E, Loh KP, Magnuson A, Flannery MA, Obrecht S, Gilmore N, Ramsdale E, Dunne RF, Wildes T, Plumb S, Patil A, Wells M, Lowenstein L, Janelsins M, Mustian K, Hopkins JO, Berenberg J, Anthony N, Dale W. Evaluation of geriatric assessment and management on the toxic effects of cancer treatment (GAP70+): a cluster-randomised study. Lancet. 2021 Nov 20;398(10314):1894-1904. doi: 10.1016/S0140-6736(21)01789-X. Epub 2021 Nov 3. PMID 34741815
- [Derived] Mohamed MR, Kyi K, Mohile SG, Xu H, Culakova E, Loh KP, Flannery M, Obrecht S, Ramsdale E, Patil A, Dunne RF, DiGiovanni G, Hezel A, Burnette B, Desai N, Giguere J, Magnuson A. Prevalence of and factors associated with treatment modification at first cycle in older adults with advanced cancer receiving palliative treatment. J Geriatr Oncol. 2021 Nov;12(8):1208-1213. doi: 10.1016/j.jgo.2021.06.007. Epub 2021 Jul 14. PMID 34272204

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 823 patients were screened. 66 failed screening and 24 withdrew before starting the intervention
Units Other Than Participants: Practice Clusters
Period: Overall Study
Arm/Group | Arm I (GA Intervention) | Arm II (Usual Care)
Started | 362; 16 Practice Clusters | 371; 24 Practice Clusters
Completed | 210; 16 Practice Clusters | 242; 24 Practice Clusters
Not Completed | 152; 0 Practice Clusters | 129; 0 Practice Clusters
Not completed — Protocol Violation | 13 | 2
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Death | 94 | 90
Not completed — Subject passively continued participation only with data obtained from their medical records | 35 | 32

BASELINE CHARACTERISTICS:
Population: There were 15 protocol violations, 13 in Arm I and 2 in Arm II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (GA Intervention) | Arm II (Usual Care) | Total
Number analyzed (Participants) | 349 | 369 | 718
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 patients did not report age, 1 from each arm.
  years
    number analyzed (Participants) | 348 | 368 | 716
    (all) | 77.2 (5.7) | 77.2 (5.2) | 77.2 (5.4)
Age, Customized [Count of Participants; unit: Participants] — Population: 2 patients did not report age, 1 from each arm.
  Participants
    Patient categorical age: number analyzed (Participants) | 348 | 368 | 716
    Patient categorical age: 70-79 years old | 244 | 250 | 494
    Patient categorical age: 80-89 years old | 94 | 110 | 204
    Patient categorical age: 90+ years old | 10 | 8 | 18
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 patients did not report sex, 1 from each arm.
  Participants
    number analyzed (Participants) | 348 | 368 | 716
    Female | 145 | 166 | 311
    Male | 203 | 202 | 405
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 341 | 365 | 706
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 12 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 40 | 12 | 52
  White | 285 | 350 | 635
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Study-reported Race/Ethnicity: Non-Hispanic White | 281 | 347 | 628
  Study-reported Race/Ethnicity: Black | 40 | 12 | 52
  Study-reported Race/Ethnicity: Other | 26 | 9 | 35
  Study-reported Race/Ethnicity: Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 349 | 369 | 718
Marital Status [Count of Participants; unit: Participants]
  Single or Never Married | 11 | 6 | 17
  Married or Domestic Partnership | 212 | 237 | 449
  Separated, Widowed, or Divorced | 125 | 125 | 250
  Unknown or Not Reported | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  Less than high school | 58 | 53 | 111
  High school graduate | 119 | 125 | 244
  Some college or above | 171 | 190 | 361
  Unknown or Not Reported | 1 | 1 | 2
Income [Count of Participants; unit: Participants]
  Less than or equal to $50,000 | 189 | 182 | 371
  More than $50,000 | 94 | 96 | 190
  Declined to answer | 65 | 90 | 155
  Unknown or Not Reported | 1 | 1 | 2
Cancer Type [Count of Participants; unit: Participants]
  Breast | 19 | 37 | 56
  Gastrointestinal | 132 | 115 | 247
  Genitourinary | 56 | 53 | 109
  Gynaecological | 29 | 14 | 43
  Lung | 64 | 116 | 180
  Lymphoma | 23 | 23 | 46
  Other | 26 | 11 | 37
Cancer Stage [Count of Participants; unit: Participants] — A diagnosis of advanced solid, incurable stage III or IV cancer was part of the eligibility criteria. Clinical staging without pathological confirmation of advanced disease was allowed. Cancer stage was collected on the "Tumor & Treatment Characteristics" measure, which is completed at baseline by the clinical research associate under the direction of the oncology physician.
  Participants
    Stage III | 42 | 35 | 77
    Stage IV | 304 | 324 | 628
    Other | 3 | 10 | 13
Previous Chemo [Count of Participants; unit: Participants] — Patient received chemotherapy before enrollment.
  Participants
    Yes | 104 | 81 | 185
    No | 234 | 277 | 511
    Unknown or Not Reported | 11 | 11 | 22
Treatment Type [Count of Participants; unit: Participants] — Type of cancer treatment the patient received. Chemotherapy is defined as cytotoxic drugs. Other agents (e.g., monoclonal antibodies and targeted agents) that have a prevalence of grade 3-5 toxicity in older patients similar to chemotherapy (>50%) were also eligible.
  Participants
    Single agent chemotherapy | 79 | 68 | 147
    Multiple agent chemotherapy | 141 | 194 | 335
    Chemotherapy and other agents | 85 | 66 | 151
    Non-chemotherapy | 44 | 41 | 85
Number GA [Mean (Standard Deviation); unit: Impairments] — There are 8 different GA domains in which impairments are measured; they include psychological status, cognition, social support, functional status, nutrition, comorbidity, polypharmacy, and physical performance. The total number of GA-domain impairments were calculated. The total number of possible impairments range from 1-8 (patients had to have at least 1 GA impairment to be eligible for the study).
  Impairments | 4.6 (1.6) | 4.4 (1.5) | 4.5 (1.6)
Number of Practice Sites [Number; unit: practice sites] | 16 | 24 | 40

OUTCOME MEASURES:

1. Primary Outcome: Patient Experienced Any Grade 3-5 Toxicity
Description: Proportion of patients who experienced grade 3-5 toxicity within 3 months of initiation of new treatment regimen. Toxicity was graded according to the National Cancer Institute (NCI) CTCAE version (v)4.0.
Time Frame: 3 months
Population: All patients who had data collected at baseline were included in this analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Arm I (GA Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 349 | 369
proportion of participants | 0.51 | 0.71
Statistical Analysis 1: Comparison: Arm I (GA Intervention) vs Arm II (Usual Care); Test type: Superiority; p = 0.0001, Mixed Models Analysis; Generalized Linear Mixed Model; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.64 to 0.86]

2. Secondary Outcome: Patient Survival at 6 Months
Description: Proportion of patients who were alive at 6 months (183 days) after enrollment estimated by Kaplan-Meier method.
Time Frame: 6 months
Population: All patients who had data collected at baseline were included in this analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Arm I (GA Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 349 | 369
proportion of participants | 0.71 | 0.74
Statistical Analysis 1: Comparison: Arm I (GA Intervention) vs Arm II (Usual Care); Test type: Superiority; p = 0.39, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.85 to 1.50]

3. Secondary Outcome: Reduced Dose Intensity
Description: Proportion of patients with reduced dose intensity in cycle 1.
Time Frame: 4-6 weeks
Population: All patients who had data collected at baseline were included in this analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Arm I (GA Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 349 | 369
proportion of participants | 0.49 | 0.35
Statistical Analysis 1: Comparison: Arm I (GA Intervention) vs Arm II (Usual Care); Test type: Superiority; p = 0.015, Mixed Models Analysis; Generalized Linear Mixed Model; Risk Ratio (RR) = 1.38, 95% CI 2-sided [1.06 to 1.78]

4. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Physical Performance.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired physical performance and starting a new treatment regimen for advanced cancer. Physical Performance measures included: Timed Up and Go, Short Physical Performance Battery, Falls History, and OARS Physical Health.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Physical Performance
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 314
Participants
  Refer to: physical therapist (outpatient or home-based depending on eligibility for home care) | 74
  Refer to: occupational therapist | 35
  Refer to: aide services | 45
  Refer to: personal emergency response information | 62
  Refer to: vision specialist if difficulties | 38
  Physical Examination: check orthostatic blood pressure | 92
  Physical Examination: decrease/eliminate blood pressure meds if blood pressure is low or low normal | 67
  Medication Review: minimize psychoactive meds including those used for supportive care | 115
  Medication Review: minimize duplicative medications | 150
  Treatment modification: consider single agent rather than doublet therapy if appropriate | 105
  Treatment modification: modify dosage | 147
  Treatment modification: modify treatment regimen | 155
  Treatment modification: conduct frequent toxicity check (weekly or every other week) | 270
  Treatment modification: choose non-neurotoxic regimen for treatment over a neurotoxic regimen | 116
  Inform: provide fall counselling handout | 270
  Inform: provide energy conservation handout | 259
  Inform: exercise or exercise prescription | 262

5. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Functional Status.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired functional status and starting a new treatment regimen for advanced cancer. Functional Status measures included: Activities of Daily Living and Instrumental Activities of Daily Living.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Functional Status
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 200
Participants
  Refer to: occupational therapist | 26
  Refer to: aide services | 32
  Refer to: personal emergency response information | 45
  Refer to: home nursing services | 25
  Physical Examination: check orthostatic blood pressure | 56
  Physical Examination: decrease/eliminate blood pressure meds if blood pressure is low or low normal | 40
  Medication Review: minimize psychoactive meds including those used for supportive care | 74
  Medication Review: minimize duplicative medications | 103
  Treatment modification: consider single agent rather than doublet therapy if appropriate | 72
  Treatment modification: modify dosage | 98
  Treatment modification: modify treatment regimen | 106
  Treatment modification: conduct frequent toxicity check | 173
  Inform: provide fall counselling handout | 170
  Inform: provide energy conservation handout | 162
  Inform: exercise or exercise prescription | 169

6. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Comorbidities.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired comorbidities and starting a new treatment regimen for advanced cancer. Comorbidity measure included: OARS Comorbidity.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Comorbidities
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 236
Participants
  Initiate direct communication with patient's primary care physician about the cancer treatment plan | 201
  Modify treatment choices: diabetes history- avoid neurotoxic agents if another option is equivalent | 45
  Modify treatment choices: heart failure history - minimize volume/infusion rate of agents | 28
  Modify treatment choices: renal impairment history - adjust as appropriate | 45
  Modify treatment choices: Modify dosage/schedule if concern about tolerance/worsening comorbidities | 113
  Provide smoking cessation counseling if the patient currently smokes | 10

7. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Cognition.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired cognition and starting a new treatment regimen for advanced cancer. Cognition measures included: Blessed Orientation Memory Concentration and Mini Cog assessments.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Cognition
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 140
Participants
  Assess decision-making capacity and if lacking elicit health care proxy information and input | 88
  Refer to: clinician experienced in memory care | 10
  Refer to: social work | 43
  Refer to: palliative care | 22
  Nueropsychological testing if dementia is suspected | 6
  TSH if dementia is suspected | 12
  B12 if dementia is suspected | 12
  Brain imaging | 16
  Provide information on cognitive rehabilitation or memory care programs | 30
  Give patient/family member handout on delirium risk | 32
  Provide explicit and written instructions for appointments, medications, and treatment | 104
  Pillbox: confirm that someone else will help fill | 62
  Pillbox: separate by am, noon, pm, and night | 53
  Medication review: minimize psychoactive and high risk medications | 89
  Treatment modification: modify treatment choice | 42
  Treatment modification: modify dosage | 68
  Treatment modification: modify treatment regimen | 61

8. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Nutrition.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired nutrition and starting a new treatment regimen for advanced cancer. Nutrition measures included: Body Mass Index, Weight Loss, and Mini Nutrition Assessment.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Nutrition
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 211
Participants
  Refer to: nutritionist/clinical dietician | 93
  Refer to: meals-on-wheels | 13
  Refer to: dentist if poor dentition or denture issues | 20
  Refer to: speech and swallow if difficulty with swallowing | 10
  Inform: nutrition handout | 169
  Treatment modification: use caution with highly emetogenic regimens and use another if appropriate | 135
  Treatment modification: utilize aggressive anti-emetic therapy | 153
  Treatment modification: conduct frequent toxicity check | 192
  Inform: mucositis handout | 133
  Recommend saline-peroxide mouthwash if treatment has high risk of mucositis | 88

9. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Social Support.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired social support and starting a new treatment regimen for advanced cancer. Social Support measure included: OARS Medical Social Support.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Social Support
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 111
Participants
  Confirm documented health care proxy is in medical record | 78
  Modify treatment choice and/or dosage | 67
  Refer or inform: ride assistance program | 22
  Refer or inform: social worker via on-site or visiting nurse services | 51
  Refer of inform: social worker via online services | 0
  Refer or inform: visiting nurse service or home health aide (if meets criteria) | 17
  Refer or inform: alternative living environments | 0
  Refer or inform: assistance programs | 0
  Refer or inform: medical insurance advising, advocacy, and negotiation | 19
  Refer or inform: legal assistance for economic and social needs | 6
  Refer or inform: community resource mobilization | 28

10. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Polypharmacy.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired polypharmacy and starting a new treatment regimen for advanced cancer. Polypharmacy measure included: medication review.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Polypharmacy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 287
Participants
  Ask patient to bring in prescribed, OTC medications, and supplements to review at the next visit | 158
  Contact primary care provider to help reduce regimen complexity | 82
  Reduce medicines solely used for hypertension or diabetes if appropriate | 59
  Consult the pharmacist to synchronize medication refills | 52
  Have pharmacist meet with the patient to evaluate drug interactions and medication counseling | 59
  Provide written instructions for taking new medications | 184
  Recommend pillbox and/or medication calendar | 123
  Provide handout on polypharmacy | 223

11. Secondary Outcome: GA-driven Recommendations Made Among Patients With Impaired Psychological Status.
Description: The type and frequency of GA-driven recommendations implemented for older patients with impaired psychological status and starting a new treatment regimen for advanced cancer. Psychological measures included: Geriatric Depression Scale and Generalized Anxiety Disorder - 7 item scale.
Time Frame: Baseline
Population: Enrolled patients in Arm 1: GA Intervention with Impaired Psychological Status
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (GA Intervention)
Number analyzed (Participants) | 107
Participants
  Provide written or verbal communication with primary care physician | 44
  Refer to: counseling or psychotherapy | 20
  Refer to: social work | 42
  Refer to: spiritual counseling or Chaplaincy services | 18
  Refer to: psychiatry if severe symptoms or if already on medications which are not adequate | 11
  Refer to: palliative care if other physical and/or cancer symptoms are present | 24
  Initiate pharmacologic therapy if appropriate in conjunction with primary care provider | 18
  Provide linkage to community resources | 30

ADVERSE EVENTS:
Time Frame: 6 months
Description: Numbers reported in this section account for all patients who had documented date of death within 183 days from the study enrollment. Note that there were 15 protocol violations, 13 in Arm I and 2 in Arm II, and these patients are not included in the at risk group.
Arm/Group | Arm I (GA Intervention) | Arm II (Usual Care)
All-Cause Mortality (participants affected / at risk) | 99/349 | 94/369
Serious Adverse Events (participants affected / at risk) | 0/349 | 0/369
Other Adverse Events (participants affected / at risk) | 0/349 | 0/369

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02054741/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT02054741/ICF_001.pdf